CLINICAL TRIAL: NCT00023790
Title: Phase I Trial of PC 4-PDT (NSC 676418) for Cutaneous Malignancies
Brief Title: Photodynamic Therapy in Treating Patients With Skin Cancer or Solid Tumors Metastatic to the Skin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1Y97; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-1Y97 (Other: Case Comprehensive Cancer Center); NCI-T99-0007; CASE-1Y97 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer; Head and Neck Cancer; Lymphoma; Metastatic Cancer; Non-melanomatous Skin Cancer; Sarcoma
Keywords: stage IV breast cancer; recurrent breast cancer; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; basal cell carcinoma of the skin; squamous cell carcinoma of the skin; recurrent skin cancer; classic Kaposi sarcoma; immunosuppressive treatment related Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; skin metastases; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Lymphoma; Neoplasm Metastasis; Sarcoma; Lymphoma, T-Cell, Cutaneous; Carcinoma, Basal Cell; Skin Neoplasms; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Mycosis Fungoides; Sezary Syndrome; Breast Neoplasms, Male | interventions — SUB1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: silicon phthalocyanine 4 — Patients receive silicon phthalocyanine 4 (Pc 4) IV over 2 hours on day 1 followed by light therapy over 30-60 minutes on day 2. Treatment repeats in 6 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of Pc 4.
  Other Names: Pc-4 (Silicone phthalocyanine)

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. This may be effective treatment for skin cancer and cancer that is metastatic to the skin.

PURPOSE: Phase I trial to study the effectiveness of photodynamic therapy in treating patients who have either squamous cell or basal cell carcinoma of the skin or solid tumors metastatic to the skin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of silicon phthalocyanine 4 (Pc 4) when administered with a fixed dose of light in patients with advanced cutaneous malignancies.
* Determine the MTD of the light when administered with a fixed dose of study drug in these patients.
* Determine the pharmacokinetics of Pc 4 in these patients.
* Determine the clinical antitumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive silicon phthalocyanine 4 (Pc 4) IV over 2 hours on day 1 followed by light therapy over 30-60 minutes on day 2. Treatment repeats in 6 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of Pc 4 and a fixed dose of light until the maximum tolerated dose (MTD) of Pc 4 is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD for Pc 4 is determined, additional patients are treated with a fixed dose of Pc 4 (2 dose levels below the MTD) and escalating doses of light until the MTD is determined. The MTD of light is defined as above.

Patients are followed at 6 weeks (or 8 weeks if treated lesion on lower extremity has not healed) and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 25-30 patients will be accrued for this study annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed tumor for which no potential curative therapy exists (e.g., surgery, radiotherapy, or systemic chemotherapy)

  * The following tumor types are eligible:

    * Cutaneous nodular metastatic breast carcinoma lesion with loco-regional cutaneous, soft tissue, or chest wall involvement

      * No chest wall recurrence without prior radiotherapy
      * Other metastatic sites allowed provided patient is concurrently receiving hormonal therapy or trastuzumab (Herceptin) of at least 4 weeks duration
    * Cutaneous or superficial subcutaneous nodular metastatic head and neck lesion
    * Cutaneous nodular Kaposi's sarcoma lesion
    * Stage IA-IIB or IVA cutaneous T-cell lymphoma (CTCL)

      * CTCL patches, plaques, or tumors with a surface area of up to 25 cm^2 if other areas of involved skin are blocked from therapy
    * Squamous cell or basal cell carcinoma of the skin that is not eligible for standard therapy (e.g., cryosurgery, radiotherapy, electrodesiccation and curettage, or excision)
    * Cutaneous and subcutaneous metastasis from any solid tumor (e.g., thoracic, gastrointestinal, or genitourinary cancers or sarcomas)
* Bidimensionally measurable disease

  * No more than 2 lesions may be treated
* No single area greater than 36 cm^2 may be treated (maximum of 25 cm^2 tumor mass with a 1 cm margin)
* Tumor treatable by surface (non-contact) light illumination
* Skin type I-III
* No tumors of the eyelids
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* No history of hepatic cirrhosis
* No hepatic disease requiring therapy

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min
* No renal disease requiring therapy

Cardiovascular:

* No myocardial infarction within the past 6 months
* No significant congestive heart failure requiring therapy
* No peripheral vascular disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Antinuclear antibody negative
* No sepsis
* No prior allergic or hypersensitivity reaction to paclitaxel vehicle
* No known photosensitivity diseases such as porphyria, systemic lupus erythematosus, xeroderma pigmentosum, or polymorphous light eruption
* No symptomatic collagen vascular disease
* Insulin-dependent or adult-onset diabetes mellitus allowed provided there are no lower extremity lesions

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior systemic chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior ultraviolet B light therapy or psoralen-ultraviolet light therapy to non-study lesions/areas
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 5 days since prior warfarin
* At least 4 weeks since prior investigational drugs
* At least 4 weeks since prior local therapy to study lesions
* At least 6 months since prior photodynamic therapy
* No concurrent aspirin, aspirin-containing medications, or non-steroidal anti-inflammatory drugs (e.g., ibuprofen, indomethacin, or cyclo-oxygenase [COX]-1 and COX-2 inhibitors)
* No other concurrent photosensitizing medications such as tetracyclines, psoralens, nalidixic acid, griseofulvin, sulfa drugs, hydrochlorothiazide, furosemide, phenothiazines, or amiodarone
* No concurrent therapeutic dosages of warfarin (non-therapeutic dosages allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-08; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by physical exam and laboratory data. | weekly for 4 weeks and in week 6
Disease response as measured by skin assessment and photography | weekly for 4 weeks and in week 6

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=cwru1y97